CLINICAL TRIAL: NCT04387019
Title: Relation Between Plasma Vitamin K2 and Glycemic Control and Metabolic Parameters in Type 2 Diabetic Patients.
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Youssry Helmy, lecturer of internal medicine ., Cairo University
Other Study IDs: N-3-2020
Record Dates: First submitted 2020-05-06; First posted 2020-05-13 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Vitamin k2 in Type 2 DM
Keywords: vitamin k2; type 2 DM; glycemic control
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — Laboratory investigations : in the form of fasting blood glucose (FBG), 2 hr postprandial blood glucose (2 hr -PPG), fasting lipids {total cholesterol (TC), triglycerides (TAG), low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C)}, glycosylated hemoglobin (Hb A1c) and Vitamin K 2 levels will be assessed .
  laboratory methodology: Two milliliters of peripheral venous blood were collected after 8 hour fasting from each participant. The measurement of Vit K2 was achieved by commercial ELISA kit based on its protocol (Glory science Co., Ltd: U.S.A.).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- I: 30 with uncontrolled type 2 DM patients
  Interventions: Diagnostic Test: blood sampling
- II: 30 controlled type 2 DM patients
  Interventions: Diagnostic Test: blood sampling
- III: 30 healthy subjects as a control group
  Interventions: Diagnostic Test: blood sampling

INTERVENTIONS:
Diagnostic Test: blood sampling — blood sampling from peripheral vein

SUMMARY:
Background and Rationale:

The agents inducing type 2 diabetes are yet to be clarified. Current studies show that several genetic and environmental parameters are associated with type 2 diabetes . Vitamin K is emerging as an important micronutrient for its beneficial role in improving insulin sensitivity and glucose metabolism and reducing the risk of type 2 diabetes (T2 D) . Studies demonstrated the lowest prevalence of Metabolic syndrome and its five components among individuals with the highest phylloquinone intake.

Objectives : The aim of our study was to evaluate the relation between plasma vitamin K2 and uncontrolled Type 2 diabetic patients.

DETAILED DESCRIPTION:
The frequency of diabetes mellitus is increasing globally and it is expected that this latent disorder will affect 300 million by 2025. Type 2 diabetes mellitus (T2DM) is a metabolic and chronic disease characterized by hyperglycemia representing the major cause of various micro and macrovascular complications

The agents inducing type 2 diabetes are yet to be clarified; however, it has been suggested that diabetes is an immune-dependent disease . Current studies show that several genetic and environmental parameters are associated with type 2 diabetes .

Vitamin K is a fat soluble vitamin . Two vitamin K- dependent-proteins, osteocalcin and matrix gamma carboxy glutamate (Gla ) protein, present in skeletal and vascular system , vitamin K exists mainly in two biologically active forms: vitamin K1 (also known as phylloquinone) and vitamin K2 (also known as menaquinone) .

According to current studies, vitamin K2 has a wider range of effects besides coagulation and functioning as a cofactor for γ--glutamate carboxylase (GGCX ) . The effect on bone is to prevent and treat osteoporosis and the effect on the cardiovascular system is to prevent and treat vascular calcification.

study by Sogabe N et al ., reported an important role of vitamin K in the regulation of dyslipidemia and vitamin K2 treatment delayed the progression of atherosclerotic plaque formation, intima-thickening, and pulmonary atherosclerosis.

study by Dam V et al ., demonstrated the lowest prevalence of Metabolic syndrome and its five components among individuals with the highest phylloquinone intake. Among the five components of Metabolic syndrome , an increase in dietary phylloquinone intake was significantly associated with a decrease in the prevalence of elevated blood pressure and reduced HDL cholesterol .

Vitamin K is emerging as an important micronutrient for its beneficial role in improving insulin sensitivity and glucose metabolism and reducing the risk of type 2 diabetes (T2 D) .

The effect of vitamin K supplementation on insulin sensitivity and glycemic status has been reviewed by study by Manna et al . They integrated currently available evidences and proposed that both vitamin K1 and vitamin K2 supplementation were beneficial to the reduced risk of T2DM. This also suggests a beneficial role of vitamin K2 on insulin sensitivity and glucose metabolism.

studies by (Yan Li et al ., 2018 - Prasenjit Manna And Jatin Kalita , 2016 ) provided an overview of the currently available studies to assess the effect of vitamin K2 supplementation on insulin sensitivity, glycaemic control and reviewed the underlying mechanisms. Overall, carboxylation of vitamin K-dependent protein osteocalcin, anti-inflammatory property, regulation of adipokine levels and lipid-lowering effect were three mechanisms underlying vitamin K2 reduced risk of T2DM and vitamin K2 had a better effect than vitamin K1 on T2DM. The interpretation of this review will increase comprehension of the development of a therapeutic strategy to prevent and treat T2DM.

Objectives:

The aim of our study was to evaluate the relation between plasma vitamin K2 and uncontrolled Type 2 diabetic patients.

Patients and methods:

A case control study including 90 subjects aged 20 to 65 years, 30 healthy subjects as a control group and 60 patients with type 2 DM .Patients will be collected from the endocrinology outpatient clinic, Kasr El Ainy, Cairo university. Patients will be divided into 3 groups, (group I) 30 patients with uncontrolled type 2 DM, (group II) 30 controlled type 2 DM and (group III) 30 non DM as control group.

All subjects will be consented and then subjected to full history taking emphasizing on the age , duration of diabetes mellitus and its treatment and full clinical examination including blood pressure measurement, weight, height, BMI (kg/m2) and waist circumference .

Laboratory investigations : in the form of fasting blood glucose (FBG), 2 hr postprandial blood glucose (2 hr -PPG), fasting lipids {total cholesterol (TC), triglycerides (TAG), low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C)}, glycosylated hemoglobin (Hb A1c) and Vitamin K 2 levels will be assessed .

laboratory methodology: Two milliliters of peripheral venous blood were collected after 8 hour fasting from each participant. The measurement of Vit K2 was achieved by commercial ELISA kit based on its protocol (Glory science Co., Ltd: U.S.A.).

-Study outcomes:

Primary outcomes :

1. Relation between plasma vitamin K2 and glycemic control in Type 2 diabetic patients.
2. Relation between plasma vitamin K2 and metabolic parameters in Type 2 diabetic patients.

Secondary outcome parameters :

1. Relation between plasma vitamin K2 and disease duration in Type 2 diabetic patients.
2. Relation between plasma vitamin K2 and forum of antidiabetic treatment in Type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 20 to 65 years old with controlled and uncontrolled DM .

Exclusion Criteria:

* • Subjects with hepatic , gastrointestinal or cardiovascular disease

  * Subjects with osteoporosis.
  * Subjects using vitamin supplements containing vitamin K.
  * Subjects using oral anticoagulants.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - 90 subjects, 60 subjects with type 2 diabetes divided into 30 with uncontrolled type 2 DM patients (group I) and 30 controlled type 2 DM patients (group II) and 30 healthy subjects as a control group (group III).
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
plasma vitamin k2 level | 3 months
  Plasma vitamin K2 level as ng/ml in type 2 diabetes patients

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No
donot share

REFERENCES:
- [Background] o Beulens JW, van der A DL, Grobbee DE et al ., ( 2010 ) . Dietary phylloquinone and menaquinones intakes and risk of type 2 diabetes. Diabetes Care 2010;33:1699-705. o Beulens, Joline WJ, Van Der A, et al ( 2010 ) . Dietary Phylloquinone and Menaquinones Intakes and Risk of Type 2 Diabetes. Diabetes Care. 2010;33:1699-705. o Cruz M, Maldonado-Bernal C, Mondragon-Gonzalez R et al., (2008) .Glycine treatment decreases proinflammatory cytokines and increases interferon-gamma in patients with type 2 diabetes. J Endocrinol Invest.;31:694-699. o Da Silva MS and Rudkowska I ( 2015 ) . Dairy nutrients and their effect on inflammatory profile in molecular studies. Mol Nutr Food Res 2015;59:1249-63. o Dam V, Dalmeijer GW, Vermeer C et al., ( 2015 ) . Association between vitamin k and the metabolic syndromea 10-year follow-up study in adults. J Clin Endocrinol Metab 2015;100:2472-9.